CLINICAL TRIAL: NCT05057208
Title: "Change of COVID-19 Vaccination Rate According to the Education, Income, Culture Level, Social Mindfulness and Prosociality "
Brief Title: Does the COVID-19 Vaccination Rate Change According to the Education, Income, Culture Level, Prosociality ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Beyza Cengiz, Medical Doctor, Pharmacology Department, Ankara University
Other Study IDs: Biophysics HacettepeUniversity
Record Dates: First submitted 2021-09-24; First posted 2021-09-27 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Vaccination Refusal
Keywords: COVID-19; Vaccination; Education level; Social mindfulness; Prosociality
MeSH Terms: conditions — Vaccination Refusal; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated: COVID Vaccinated
  Interventions: Biological: COVID
- Non-vaccinated: COVID Non-vaccinated

INTERVENTIONS:
Biological: COVID — COVID vaccination
  Groups: Vaccinated

SUMMARY:
"Does the COVID-19 vaccination rate change according to the education, income, culture level, social mindfulness and prosociality ?"

DETAILED DESCRIPTION:
In this study the investigators will examine the correlation of the COVID-19 vaccination rates of the cities with income, cultural level and various education levels. Furthermore, vaccination rate change with respect to social mindfulness and prosociality will be investigated also? The investigators hypothesize that a) Income & culture level is positively correlated with vaccination rate, b) If "time spent in education" increases (from illiterate, primary/mid/high school to BSc, MSc & PhD) vaccination level increases, c) if social mindfullness or prosociality increases, vaccination rate increase also? The results of this study make it easier for us to understand why anti-vaccine people are against vaccination. The results may lead to more different variables and questions being included in questionnaires to understand resistance against vaccination.

Our basic variables are vaccination rates of cities, education level distribution (illiterate, primary school, middle school, high school, bachelor's degree, master degree, doctoral degree percentages) of cities, per capita income in the city, number of movie theaters per capita in the city and internet book sales of cities in Turkey. the investigators will do this work for other countries also as new data become available.

For social mindfulness and prosociality vs. vaccination rate investigation, the investigators will use primarily Doesum et al.'s 2021 research variables: SVO (Social value orientation) and SoMi (Social Mindfulness) with WHO vaccination rate tables.

ELIGIBILITY:
Inclusion Criteria:

* over 15 years old

Exclusion Criteria:

* under 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals over the age of 15 in Turkey 31 countries with SVO and SoMi index
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Change of Vaccination Rate | 8 months
  Our basic variables are vaccination rates of cities, education level distribution (illiterate, primary school, middle school, high school, bachelor's degree, master degree, doctoral degree percentages) of cities, per capita income in the city, number of movie theaters per capita in the city and internet book sales of cities in Turkey and SVO (Social value orientation) and SoMi (Social Mindfulness) in different countries with WHO vaccination rate tables. The results of this study make it easier for us to understand why anti-vaccine people are against vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In 8 months, the investigators will calculate correlation of variables(Education, income, culture level, social mindfulness and prosociality)

REFERENCES:
- [Background] Van Doesum NJ, Murphy RO, Gallucci M, Aharonov-Majar E, Athenstaedt U, Au WT, Bai L, Bohm R, Bovina I, Buchan NR, Chen XP, Dumont KB, Engelmann JB, Eriksson K, Euh H, Fiedler S, Friesen J, Gachter S, Garcia C, Gonzalez R, Graf S, Growiec K, Guimond S, Hrebickova M, Immer-Bernold E, Joireman J, Karagonlar G, Kawakami K, Kiyonari T, Kou Y, Kuhlman DM, Kyrtsis AA, Lay S, Leonardelli GJ, Li NP, Li Y, Maciejovsky B, Manesi Z, Mashuri A, Mok A, Moser KS, Motak L, Netedu A, Pammi C, Platow MJ, Raczka-Winkler K, Reinders Folmer CP, Reyna C, Romano A, Shalvi S, Simao C, Stivers AW, Strimling P, Tsirbas Y, Utz S, van der Meij L, Waldzus S, Wang Y, Weber B, Weisel O, Wildschut T, Winter F, Wu J, Yong JC, Van Lange PAM. Social mindfulness and prosociality vary across the globe. Proc Natl Acad Sci U S A. 2021 Aug 31;118(35):e2023846118. doi: 10.1073/pnas.2023846118. PMID 34426492
- See also: Vaccination rate in countries — https://ourworldindata.org/covid-vaccinations?country=OWID_WRL